CLINICAL TRIAL: NCT00833261
Title: A Phase II Multi-Center Study of Concomitant Cetuximab and Cisplatin With Re-Irradiation Using Intensity-Modulated Radiotherapy in Patients With Recurrent Squamous Cell Carcinoma of the Head-and-Neck
Brief Title: Nab-Paclitaxel, Cetuximab, Cisplatin, and Radiation Therapy in Treating Patients With Recurrent Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000632295; SCCC-04308; CA 225314; 112008-004
Record Dates: First submitted 2009-01-30; First posted 2009-02-02 (Estimated); Results first posted 2019-07-05 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2018-11

CONDITIONS: Head and Neck Cancer
Keywords: recurrent hypopharynx Cancer; recurrent larynx Cancer; recurrent verrucous carcinoma; squamous cell carcinoma; recurrent oral cavity cancer; recurrent metastatic occult primary cancer; recurrent oropharynx cacner; recurrent paranasal sinus and nasal cavity cancer; tongue cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Hypopharyngeal Neoplasms; Laryngeal Neoplasms; Carcinoma, Verrucous; Carcinoma, Squamous Cell; Mouth Neoplasms; Tongue Neoplasms | interventions — Cetuximab; Drug Therapy; Cisplatin; Radiotherapy, Intensity-Modulated; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm: Chemotherapy with Concurrent Radiation therapy (Experimental): Nab-Paclitaxel, Cetuximab, Cisplatin, and Radiation Therapy intensity-modulated radiation therapy
  Interventions: Drug: cetuximab; Drug: cisplatin; Radiation: intensity-modulated radiation therapy; Drug: Nab-Paclitaxel

INTERVENTIONS:
Drug: cetuximab — cetuximab
  Other Names: chemo
Drug: cisplatin — cisplatin
  Other Names: chemo
Radiation: intensity-modulated radiation therapy — IMRT
  Other Names: IMRT
Drug: Nab-Paclitaxel — Nab-Paclitaxel
  Other Names: chemo

SUMMARY:
RATIONALE: Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Drugs used in chemotherapy, such as cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving cetuximab and cisplatin together with radiation therapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving cetuximab and cisplatin together with radiation therapy works in treating patients with recurrent head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate whether treatment with cetuximab, cisplatin, and intensity-modulated radiotherapy improves the overall survival of patients with recurrent squamous cell carcinoma of the head and neck.

Secondary

* To determine the progression-free survival and local-regional progression in these patients.
* To identify and estimate the incidence rate of acute and late toxicities associated with this treatment regimen.
* To determine the pattern of disease progression in these patients.

OUTLINE: This is a multicenter study.

Patients receive cetuximab IV over 60-120 minutes once weekly in weeks 1-7. Patients also receive cisplatin IV over 60 minutes once weekly and undergo intensity-modulated radiotherapy once daily 5 days a week in weeks 2-7.

After completion of study treatment, patients are followed every 3 months for 2 years and then every 6 months for 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Pathologically confirmed squamous cell carcinoma (SCC) of the upper aerodigestive tract
* Recurrent disease or second primary SCC

  * Recurrence or second primary must be confined to the head and neck above the clavicles (loco-regional recurrence)
  * Majority (≥ 75%) of the recurrent tumor must be in areas previously irradiated to ≥ 45 Gy
  * More than one recurrence allowed provided the first recurrence occurred > 6 months after the completion of prior radiotherapy
* Unresectable disease OR has high-risk features after resection (e.g., positive margins and/or extracapsular extension)

  * No signs of carotid exposure
* No primary nasopharyngeal or salivary gland tumor
* Equivocal pulmonary nodes on chest CT scan allowed provided they are < 1 cm, cannot be safely biopsied, or are negative on PET scan
* No distant metastasis

PATIENT CHARACTERISTICS:

* Karnofsky performance status 70-100%
* ANC ≥ 2,000/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 8.0 g/dL (transfusion or other intervention allowed)
* Bilirubin < 1.5 mg/dL
* AST or ALT < 2 times upper limit of normal
* Creatinine clearance ≥ 50 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Able to submit prior radiotherapy records to assure that the spinal cord tolerance is not exceeded
* No active cardiac disease, including any of the following:

  * Unstable angina
  * Uncontrolled hypertension
  * Myocardial infarction within the past 6 months (unless successfully treated with coronary artery bypass graft or percutaneous transluminal coronary angioplasty)
  * Uncontrolled arrhythmia
  * Congestive heart failure
  * At least 3 heart-related hospitalizations within the past year
* No severe chronic obstructive pulmonary disease requiring ≥ 3 hospitalizations within the past year
* No concurrent medical illness that would impair patient tolerance to therapy or limit survival
* No other invasive malignancy within the past 2 years
* No pre-existing peripheral sensory neuropathy ≥ grade 2
* No prior severe infusion reaction to a monoclonal antibody
* No prisoners or individuals who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious) illness

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from prior surgery
* Prior cisplatin and cetuximab allowed
* At least 6 months since prior radiotherapy or chemotherapy
* No prior radiotherapy > 75 Gy
* No prior chemotherapy for recurrent head and neck cancer

  * Prior chemotherapy as a component of the primary treatment allowed
* No prior combination cisplatin, cetuximab, and radiotherapy for recurrent head and neck cancer

  * Patients with a new primary head and neck cancer whose prior primary head and neck cancer was treated with concurrent cisplatin, cetuximab, and radiotherapy are eligible provided it has been > 6 months since treatment

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2008-12 (Actual); Primary Completion 2013-09 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Baylor Research Institute, Dallas, Texas
  - University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Awan MJ, Nedzi L, Wang D, Tumati V, Sumer B, Xie XJ, Smith I, Truelson J, Hughes R, Myers LL, Lavertu P, Wong S, Yao M. Final results of a multi-institutional phase II trial of reirradiation with concurrent weekly cisplatin and cetuximab for recurrent or second primary squamous cell carcinoma of the head and neck. Ann Oncol. 2018 Apr 1;29(4):998-1003. doi: 10.1093/annonc/mdy018. PMID 29346519

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm: Chemotherapy With Concurrent Radiation Therapy: Nab-Paclitaxel, Cetuximab, Cisplatin, and Intensity-modulated radiation therapy (IMRT)
Period: Overall Study
Arm/Group | Single Arm: Chemotherapy With Concurrent Radiation Therapy
Started | 37
Completed | 33 (3 patients withdrew from the study prior to treatment & 1 receiving it did not complete the course.)
Not Completed | 4
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Population: Three patients withdrew from the study prior to treatment.
Arm/Group | Single Arm: Chemotherapy With Concurrent Radiation Therapy
Number analyzed (Participants) | 34
Age, Continuous [Median (Full Range); unit: years] — Population: One patient receiving treatment did not complete the entire course of systemic therapy
  years
    number analyzed (Participants) | 33
    (all) | 55.5 [45 to 76]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One patient receiving treatment did not complete the entire course of systemic therapy
  Participants
    number analyzed (Participants) | 33
    Female | 12
    Male | 21
Region of Enrollment [Number; unit: participants] — Population: One patient receiving treatment did not complete the entire course of systemic therapy
  participants
    United States: number analyzed (Participants) | 33
    United States | 33

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: The 2-year PFS was measured from the date of enrollment to the first occurrence of new metastatic lesions, objective tumor progression, or death. The combination of cisplatin and cetuximab concurrent with radiation therapy for head and neck cancer has shown to have a favorable PFS. Patients were followed until death or from 7.5 months to 63.6 months (median 25.6 months) in those alive at last evaluation.
Time Frame: 2 year from the date of enrollment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Single Arm: Chemotherapy With Concurrent Radiation Therapy
Number analyzed (Participants) | 33
percentage of participants | 60 [42 to 78]

2. Secondary Outcome: Number of Participants With Acute and Late Toxicities
Description: Incidence rate of acute and late toxicities of grade 3 or higher was measured after each treatment cycle was over. The most common late toxicities defined as toxicity occurring more than 90 days after treatment included laryngeal edema and xerostomia.
Time Frame: 6 months within the end of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm: Chemotherapy With Concurrent Radiation Therapy
Number analyzed (Participants) | 33
Participants | 21

ADVERSE EVENTS:
Arm/Group | Single Arm: Chemotherapy With Concurrent Radiation Therapy
All-Cause Mortality (participants affected / at risk) | 0/33
Serious Adverse Events (participants affected / at risk) | 21/33
Other Adverse Events (participants affected / at risk) | 10/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm: Chemotherapy With Concurrent Radiation Therapy (N=33)
Lymphopenia (Blood and lymphatic system disorders) | 21 (21)
Leukopenia (Blood and lymphatic system disorders) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 4 (4)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Infection (Infections and infestations) | 7 (7)
Dermatitis (Injury, poisoning and procedural complications) | 6 (6)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm: Chemotherapy With Concurrent Radiation Therapy (N=33)
Anorexia (General disorders) | 5 (5)
pain (General disorders) | 10 (10)
Dysphagia (Gastrointestinal disorders) | 8 (8)
Other electrolyte abnormalities (Blood and lymphatic system disorders) | 8 (8)
Fatigue (General disorders) | 3 (3)
Hyponatremia (General disorders) | 3 (3)
Hypophosphatemia (Blood and lymphatic system disorders) | 3 (3)
Mucositis (Gastrointestinal disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes